CLINICAL TRIAL: NCT06392087
Title: Prehospital Analgesia in Adults Using Inhaled (PAIN) Methoxyflurane Study
Brief Title: Prehospital Analgesia in Adults Using Inhaled Methoxyflurane Study
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20240319100
Record Dates: First submitted 2024-03-19; First posted 2024-04-30 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pain, Acute
Keywords: paramedic; traumatic pain; Ambulance
MeSH Terms: conditions — Acute Pain | interventions — Methoxyflurane; Standard of Care

STUDY DESIGN:
Intervention Model Description: Step Wedge Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control standard care (Active Comparator): The patients who meet the indications of the study trauma-related pain Moderate/Severe (>4 verbal numeric pain score), are provided current standard of care for pain (Advil or Ketorolac/Tylenol, opioids (for Advanced Care paramedics)
  Interventions: Other: Standard Care
- Intervention (Experimental): The patients who meet the indications of the study trauma-related pain Moderate/Severe (>4 verbal numeric pain score) and receive methoxyflurane
  Interventions: Drug: Methoxyflurane

INTERVENTIONS:
Drug: Methoxyflurane — Patients ≥ 18 years of age (using a waiver of consent process) Pain score ≥ 4 on the verbal numeric pain rating scale (NPRS) traumatic injury (defined as: physical injuries of sudden onset and severity which requires immediate medical attention) Unaltered (Glasgow Coma Scale (GCS) ≥ 14) Normotensive (systolic blood pressure ≥100) Treated and transported
  Other Names: Penthrox
  Arms: Intervention
Other: Standard Care — Patients ≥ 18 years of age (using a waiver of consent process) Pain score ≥ 4 on the verbal numeric pain rating scale (NPRS) traumatic injury (defined as: physical injuries of sudden onset and severity which requires immediate medical attention) Unaltered (Glasgow Coma Scale (GCS) ≥ 14) Normotensive (systolic blood pressure ≥100) Treated and transported
  Arms: Control standard care

SUMMARY:
This study is about a new pain relief medication called methoxyflurane. Pain from injuries, like broken bones, is a big reason people call ambulances. It's important to treat pain well because it can make people sick and slow down healing. But often, pain isn't treated enough, which can lead to more problems.

Paramedics use different drugs to manage pain, but some are hard to give and need special training and equipment. Methoxyflurane is a new option. It's a gas you breathe in through a special inhaler. It's been used in Australia and New Zealand for a long time and has shown to work quickly and safely for different kinds of pain.

This study wants to see if methoxyflurane works well for people with moderate to severe pain from injuries compared to other medicines like Advil, Tylenol and opioids. It's testing if methoxyflurane can give fast pain relief and if paramedics find it easy to use. The study will help understand if methoxyflurane could be a good option for treating pain in ambulances.

DETAILED DESCRIPTION:
The aim of this multi-centred study is to evaluate the prehospital use of methoxyflurane in patients ≥ 18 years of age presenting with moderate to severe pain (verbal numeric pain rating scale (NPRS) ≥ 4) secondary to trauma (which is defined as a physical injury of sudden onset and severity which requires immediate medical attention) as compared to other current therapies available to paramedics (NSAIDS and Opioids).

This will be a prehospital prospective stepped-wedge open-label, non-blinded, cluster randomized trial, enrolling patients with trauma related moderate to severe pain (numerical pain rating scale ≥4). It will be composed of three phases, involving a total of seven Ontario paramedic services. Our 24-month study will consist of the three following phases: 1) a 6-month setup and training period, followed by phase 2) the stepped-wedge trial (8-months) and phase 3) a 9-month period for data analysis and knowledge dissemination.

The verbal numeric pain rating scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numeric scale. The scale is comprised of values ranging from 0 (no pain at all) to 10 (worst imaginable pain). After ethics approvals have been secured for all sites, and after the initial 4-week observation period (where paramedics will provide standard care) one paramedic service will be randomized, using a number generator which the study team will be blinded, to the intervention condition (Methoxyflurane). Additional paramedic services will subsequently be randomized, and notified one by one at 4 week intervals until all seven paramedic services have been randomized to the intervention arm. Data will be collected for all eligible patients in each paramedic service for a total duration of 8 months. The study will be conducted in seven paramedic services in Eastern Ontario and will enrol patients who have been treated by paramedics, trained and authorized in the use and administration of methoxyflurane.

Eastern Ontario comprises 35 300 km2 and has a total regional population of 1.76 million. There are eight base hospitals in Ontario that provide medical direction, leadership and advice in the provision of prehospital emergency care. The Regional Paramedic Program for Eastern Ontario (RPPEO) is the base hospital which provides oversight to the seven included paramedic services. These paramedic services are comprised of 944 paramedics (738 of which are Primary Care Paramedics and 256 who are Advanced Care Paramedics). In summary, this study will comprise seven land paramedic services, operating in a catchment area of 10 rural counties and 4 cities, with 18 acute care hospitals and 1 university hospital.

ELIGIBILITY:
Inclusion Criteria:

Indications for analgesia therapy:

* Patients ≥ 18 years of age (using a waiver of consent process)
* Pain score ≥ 4 on the verbal numeric pain rating scale (NPRS)
* traumatic injury (defined as: physical injuries of sudden onset and severity which requires immediate medical attention)
* Unaltered (Glasgow Coma Scale (GCS) ≥ 14)
* Normotensive (systolic blood pressure ≥100)
* Treated and transported

Patients will be given methoxyflurane as soon as the treating paramedic has determined they meet inclusion criteria.

Paramedics will follow the Advanced Life Support Patient Care Standards21 for all other care the patient requires (including pain directive if methoxyflurane does not control pain after 10 min).

Contraindications listed in the ALS-PCS will be used by paramedics in providing analgesia. Within the standards paramedics are required to record vital signs every 5 minutes including verbal NPRS.

Exclusion Criteria:

Patients with the following characteristics will be excluded (based on the Health Canada Product Monograph):

* History or family history of malignant hyperthermia
* Age <18 years of age
* Pregnancy or breast-feeding
* Inclusion in another study not allowing the co-enrollment
* Known renal impairment
* Known liver disease
* History of use of methoxyflurane in the last 3 months
* Allergy to methoxyflurane

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Verbal Numeric Pain Score | 10 min
  verbal numeric pain rating score (NPRS) initial and at 10 min, 0 referring to no pain and 10 severe pain

SECONDARY OUTCOMES:
Rescue Medications | 10 min
  (as defined by addition of any other pain medication (ketorolac or opioids (fentanyl or morphine) 10 min after methoxyflurane administration, during paramedic care)
Transport Time | 8 months
  From time onscene, to hospital arrival
Time to first analgesia | 8 months
  time to first administration of analgesia (NSAIDs, Opioids or methoxyflurane)
Vital signs | 5 min
  vital signs (Blood pressure, Heart rate, oxygen saturation, temperature, respiratory rate, level of consciousness) (initial and at arrival to hospital) (repeat measures will be captured in data every 5 mins)
Verbal numeric pain score during care | 5 min
  verbal numeric pain rating score (NPRS) initial and at 10 min, 0 referring to no pain and 10 severe pain (as transport times will vary)

OTHER OUTCOMES:
Adverse events | 8 months
  adverse events post administration of analgesia: any advanced airway interventions, oxygen requirement (oxygen saturations <94%), drop in blood pressure by 40% and/or <90 systolic, complaints of nausea or vomiting, malignant hyperthermia reaction).

IPD SHARING:
Plan to Share IPD: Undecided
de-identified data will be considered if requested for sharing.